CLINICAL TRIAL: NCT07041788
Title: A Prospective, Single-Arm Clinical Trial of Iparomlimab and Tuvonralimab Combined With Spatially Fractionated Radiotherapy and Definitive Chemoradiotherapy in Locoregionally Advanced Bulky Head and Neck Squamous Cell Carcinoma
Brief Title: Iparomlimab and Tuvonralimab Combined With SFRT and Definitive Chemoradiotherapy in Locoregionally Advanced Bulky HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-I-2025-013
Record Dates: First submitted 2025-03-26; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Spatially Fractionated Radiation Therapy; Ipalontilimab and Tuvorilimab; Locoregionally advance head and neck squamous cell carcinoma
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study of Iparomlimab and Tuvonralimab Combined With SFRT and Definitive Chemoradiotherapy in HNSCC (Experimental): This is a single-arm study.(1) Induction therapy: Administer Spatially Fractionated Radiotherapy to the tumor at a dose of 10 - 20 Gy in 1 fraction. Subsequently, conduct 3 cycles of induction chemotherapy (docetaxel 75 mg/m² on day 1, cisplatin 25 mg/m² from day 1 to day 3, every 3 weeks for 3 cycles) combined with immunotherapy using Iparomlimab and Tuvonralimab (5 mg/kg on day 1, every 3 weeks for 3 cycles).
  (2) Concurrent chemoradiotherapy: Initiate radical concurrent chemoradiotherapy within 2 - 4 weeks after the completion of induction therapy. The prescribed dose of radical radiotherapy is 70 Gy for the primary tumor and 66 - 70 Gy for the positive cervical lymph nodes, to be delivered in 30 - 33 fractions. Concurrent chemotherapy involves intravenous.
  (3) Maintenance therapy: Start maintenance immunotherapy with Iparomlimab and Tuvonralimab 4 - 6 weeks after the completion of concurrent chemoradiotherapy. Administer it at a dose of 5 mg/kg per administration.
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection — Induction Therapy:
  Spatially Fractionated Radiotherapy: Administer 10-20 Gy in a single fraction to the tumor.
  Chemotherapy + Immunotherapy:
  Docetaxel 75 mg/m² IV on Day 1. Cisplatin 25 mg/m² IV on Days 1-3. Iparomlimab and Tuvonralimab Injection 5 mg/kg IV on Day 1. Cycles: Every 3 weeks (Q3W) for 3 cycles.
  Maintenance Therapy:
  Begin 4-6 weeks after radiotherapy completion.
  Iparomlimab and Tuvonralimab:
  Dose: 5 mg/kg diluted in 100 mL 0.9% NaCl or 5% glucose. Administration: IV infusion over ≥20 minutes (total duration including flushing ≤60 minutes).
  Cycles: Q3W for 14 cycles (maximum 1 year).
  Iparomlimab and Tuvonralimab Injection:
  Continue until disease progression, intolerable toxicity, initiation of new anti-tumor therapy, withdrawal of consent, or investigator decision to discontinue.
  Maximum treatment duration: 1 year.

SUMMARY:
Study Objectives

1. Primary Objective:

   The core aim of this study is to investigate whether the sequential approach of Spatially Fractionated Radiotherapy followed by 3 cycles of induction chemotherapy combined with Iparomlimab and Tuvonralimab, definitive chemoradiotherapy, and maintenance therapy with the Iparomlimab and Tuvonralimab can improve the 2-year event-free survival (EFS) rate in patients with locoregionally advanced bulky head and neck squamous cell carcinoma (HNSCC).
2. Secondary Objectives:s

To analyze the impact of this integrated treatment regimen on key efficacy endpoints, including:

Objective response rate (ORR), Duration of response (DoR), Distant metastasis-free survival (DMFS), Local region recurrence-free survival (LRRFS), Overall survival (OS)。 2. Study Endpoints

(1) Primary Endpoint and Definition: 2-Year Event-Free Survival (EFS) Rate (2) Secondary Endpoints and Definitions:

1. 2-Year Overall Survival (OS) Rate
2. 2-Year Distant Metastasis-Free Survival (DMFS) Rate.
3. 2-Year Local Region Recurrence-Free Survival (LRRFS) Rate.
4. Objective Response Rate (ORR).
5. Duration of Response (DoR).
6. Quality of Life (QoL):

   Assessed across multiple domains:

   Physical Function: Measured via tools like the 6-minute walk test or ADL (Activities of Daily Living) scale.

   Psychological Status: Evaluated using instruments such as HAMD (Hamilton Anxiety and Depression Scale) or MMSE (Mini-Mental State Examination).

   Social Function: Assessed via social engagement questionnaires (e.g., HAQ-DI [Health Assessment Questionnaire-Disability Index]).

   Spiritual Well-being: Evaluated using tools like PIL (Purpose in Life test). Clinically meaningful improvements in these domains before and after treatment define successful QoL endpoints (e.g., positive changes in physical, psychological, social, and spiritual health in cardiac patients).
7. Safety:

   The nature and severity of adverse reactions associated with the treatment.
8. Tolerability:

The degree to which patients can endure treatment-related side effects.

DETAILED DESCRIPTION:
I. Study Design and Technical Route Details 1. Stratified Implementation of Treatment Protocols

1. Spatially Fractionated Radiotherapy (SFRT) Phase Technical Parameters: Three-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiotherapy (IMRT) is used to deliver a single high-dose fraction to the primary tumor and bulky metastatic lymph nodes (≥5 cm), with a prescribed dose of 10-20Gy/1 fraction. Dose-volume histogram (DVH) optimization ensures target coverage while limiting doses to organs at risk (e.g., spinal cord ≤45Gy, parotid gland mean dose ≤26Gy).

   Timing: A positioning CT scan (slice thickness ≤3 mm) is completed within 7 days of enrollment. The radiation oncologist contours the target volumes, and the physicist designs the treatment plan, which is reviewed by a multidisciplinary team (MDT) before implementation.
2. Induction Chemotherapy Combined with Immunotherapy Phase

   Drug Regimen:

   Docetaxel: 75mg/m², intravenous drip, d1, Q3W for 3 cycles (body surface area calculated using measured height and weight, precise to 0.01m²).

   Cisplatin: 25mg/m², intravenous drip, d1-3, Q3W for 3 cycles (hydration pretreatment required, daily fluid intake ≥2000ml, electrolyte monitoring).

   Iparomlimab and Tuvonralimab: 5mg/kg, intravenous infusion, d1, Q3W for 3 cycles (diluted in 100ml 0.9% sodium chloride solution, infusion duration ≥30 minutes; electrocardiographic monitoring required for the first dose).

   Cycle Transition: Induction therapy starts within 7 days after SFRT. Each chemotherapy cycle requires confirmation of normal blood counts (ANC ≥1.5×10⁹/L, PLT ≥90×10⁹/L) and liver/kidney function (ALT/AST ≤2.5×ULN) before initiation.
3. Definitive Concurrent Chemoradiotherapy Phase

   Radiotherapy Protocol:

   Target Volume Definition: GTVₜₙ₀ (primary tumor) receives 70Gy/30-33 fractions, GTVₙ (positive lymph nodes) receives 66-70Gy/30-33 fractions, and clinical target volume (CTV) receives 54-60Gy/30-33 fractions. IMRT is used with daily fractions (2Gy/fraction), total treatment time ≤6 weeks.

   Concurrent Chemotherapy: Cisplatin 100mg/m², infused over 3 days (d1-3), Q3W for 2 cycles. Chemotherapy starts simultaneously with radiotherapy, within 48 hours of each other.
4. Immunotherapy Maintenance Phase Protocol: Iparomlimab and Tuvonralimab 5mg/kg, Q3W, intravenous infusion for 14 cycles (total treatment duration ~1 year).

Discontinuation Criteria: Disease progression (RECIST 1.1), intolerable toxicity (CTCAE ≥3), patient withdrawal of informed consent, or investigator-determined need to exit.

2. Technical Details of Efficacy Assessment

Imaging Evaluation:

Baseline Scans: Pre-enrollment head and neck contrast-enhanced CT/MRI (slice thickness ≤3 mm), chest CT, and whole-body bone scan; PET-CT as needed.

Dynamic Evaluation: Repeat scans at the end of induction therapy, 1 month after concurrent chemoradiotherapy, and every 12 weeks during follow-up. Image registration techniques ensure target reproducibility.

Biomarker Detection: Peripheral blood samples (5ml EDTA anticoagulated tubes) are collected before treatment, after induction therapy, and during maintenance therapy to detect PD-L1 expression (immunohistochemistry), T-cell subsets (flow cytometry), and 12 cytokines (ELISA, including IL-1β, IL-6, TNF-α, etc.).

II. Safety Management System

1. Adverse Event (AE) Monitoring and Management Real-Time Tracking: AEs are recorded at each visit with details on onset time, duration, severity (CTCAE 5.0 grading), and causality to treatment. Particular attention is paid to immune-related adverse events (irAEs), such as pneumonitis, colitis, and thyroid dysfunction.

   Grading Management:

   Grade 1-2 AEs: Close observation with symptomatic support as needed (e.g., antiemetics, antipyretics); no dose adjustment required.

   Grade 3 AEs: Treatment suspension until recovery to ≤Grade 1; restart with unchanged Iparomlimab/Tuvonralimab dose, while chemotherapy dose may be reduced by 20%.

   Grade 4-5 AEs or Fatal irAEs: Permanent discontinuation; multidisciplinary consultation initiated, with potential administration of glucocorticoids (e.g., methylprednisolone 1-2mg/kg/d) or immunosuppressants.
2. Special Toxicity Monitoring Hematological Toxicity: Weekly blood count monitoring during induction and concurrent chemotherapy. For ≥Grade 3 neutropenia or thrombocytopenia, G-CSF (e.g., PEG-rhG-CSF 6mg subcutaneously) or platelet transfusions are administered, with prophylactic antibiotics (e.g., levofloxacin) until ANC ≥1.0×10⁹/L.

Radiation-Induced Injury: Weekly assessment of oral mucositis (RTOG grading) and skin reactions (CTCAE) during radiotherapy. Patients receive oral rinses (e.g., chlorhexidine) and skin protectants (e.g., Biafine); severe cases require radiotherapy suspension and analgesia.

III. Data Management and Quality Control

1. Data Collection and Documentation Case Report Form (CRF): An electronic CRF (eCRF) system is used for real-time recording of baseline characteristics, treatment processes, efficacy evaluations, and AE data to ensure traceability.

   Biological Sample Management: Tumor tissue samples (surgical or biopsy specimens) and blood samples are stored at -80°C with unique identifiers. A sample tracking database records storage locations, collection times, and usage (limited to study-related testing).
2. Quality Control Measures Internal Audits: Research coordinators verify CRF data integrity weekly, with quarterly on-site audits by the institutional office focusing on treatment compliance, AE underreporting, and sample management gaps.

External Review: An independent Data Monitoring Committee (DMC) convenes annually to review safety data and efficacy endpoints. A predefined stopping rule triggers early termination if treatment-related mortality ≥2%.

IV. Ethics and Compliance

1. Ethical Review Process Initial Approval: The study protocol, informed consent form (ICF), and 附属文件 (supporting documents) must undergo review and obtain approval from the Ethics Committee of the Second Affiliated Hospital of Nanchang University before initiation.

   Protocol Amendments: Any protocol modifications (e.g., dose adjustments, inclusion/exclusion criteria) require resubmission to the Ethics Committee for review, with amendments communicated to all research staff upon approval.
2. Protection of Subject Rights Informed Consent: Principal investigators provide detailed explanations of study objectives, risks, and benefits to subjects and their families, allowing a 48-hour consideration period. Informed consent is confirmed through written signatures and audio-video recording to ensure unambiguous understanding.

Insurance Coverage: Each subject is enrolled in a clinical trial liability insurance (¥300,000 per subject), covering medical expenses and compensation for treatment-related injuries.

V. Human Genetic Resources Management Sample Usage Scope: Samples are used exclusively for study-related biomarker testing and are not provided to external parties or exported.

Destruction Procedures: Remaining samples are destroyed under dual supervision after study completion, with documentation of destruction time, quantity, and method, subject to Ethics Committee approval.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, both sexes eligible;
2. Histologically confirmed head and neck squamous cell carcinoma (HNSCC), diagnosed as locoregionally advanced disease with measurable primary tumor and/or cervical metastatic lymph nodes >5 cm in maximum diameter, and deemed unresectable by surgical evaluation;
3. Treatment-naive (no prior anti-tumor therapy);
4. At least one measurable lesion (excluding brain metastases) per RECIST 1.1 criteria;
5. ECOG performance status 0-1;
6. Life expectancy ≥12 weeks;
7. Organ function meeting the following criteria (no blood products, colony-stimulating factors, leukocyte/ thrombocyte/ erythrocyte-stimulating agents within 14 days prior to first study drug administration):

   1. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
   2. Platelets ≥90×10^9/L;
   3. Hemoglobin ≥8 g/dL;
   4. Serum albumin ≥2.8 g/dL;
   5. Total bilirubin ≤1.5×ULN, ALT/AST/ALP ≤2.5×ULN; if liver metastases present, ALT/AST ≤5×ULN; if liver/bone metastases present, ALP ≤5×ULN;
   6. Serum creatinine ≤1.5×ULN or creatinine clearance >60 mL/min;
   7. APTT and INR ≤1.5×ULN (patients on stable anticoagulation [e.g., LMWH, warfarin] with therapeutic INR acceptable for screening).
8. Voluntary informed consent, good compliance, and willingness to cooperate with follow-up;
9. Investigator determination of potential benefit.

Exclusion Criteria:

1. Those with a history of severe immediate - type allergic reactions to any of the drugs used in this study；
2. Within six months before screening, having any of the following conditions: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism. Patients known to have coronary artery disease, congestive heart failure that doesn't meet the above criteria, or a left ventricular ejection fraction of less than 50% must have an optimally stable medical regimen as determined by the treating physician. If appropriate, a cardiologist can be consulted；
3. Individuals who have received anti - tumor vaccines or live vaccines within four weeks before the first administration of the study drug；
4. Patients with active autoimmune diseases or a history of autoimmune diseases that are likely to relapse. The following patients are not excluded and can proceed to further screening:

   1. Those with well - controlled type 1 diabetes.
   2. Patients with hypothyroidism that can be controlled with hormone replacement therapy alone.
   3. People with skin diseases that do not require systemic treatment, such as vitiligo, psoriasis, and alopecia.
   4. Any other diseases that are not expected to relapse without external triggers；
5. Those lacking full or restricted civil capacity；
6. Patients with physical or mental disorders who, in the investigator's opinion, are unable to fully or adequately understand the potential complications of this study；
7. Patients with an expected survival time of less than three months；
8. Patients with significantly reduced functions of the heart, liver, lungs, kidneys, and bone marrow；
9. Those with a history of substance abuse or alcohol addiction；
10. Patients whose tumor lesions invade large blood vessels, such as the internal carotid artery and jugular vein and their main branches, with a high risk of bleeding；
11. Subjects who need systemic treatment with corticosteroids (more than 10 mg/day prednisone equivalent) or other immunosuppressants within two weeks before the first use of the study drug, except for the use of corticosteroids for local esophageal inflammation and the prevention of allergies, nausea, and vomiting. In other special cases, communication with the sponsor is required. In the absence of active autoimmune diseases, the inhalation or local use of steroids and adrenal cortical hormone replacement at a dose higher than 10 mg/day prednisone equivalent is allowed；
12. Those with a history of immunodeficiency, including HIV - positive results, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation；
13. Pregnant or lactating female patients, as well as male or female patients who are fertile but unwilling or unable to use contraception throughout the study and for at least one year after the end of the treatment plan；
14. Patients who, in the investigator's opinion, are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2028-07-09 (Estimated); Study Completion 2030-07-09 (Estimated)

PRIMARY OUTCOMES:
2-year EFS (Event - Free Survival) | 2 years
  Event-Free Survival (EFS) rate: Defined as the time from enrollment to the occurrence of the first event among any of the following: disease progression (including local progression and distant metastasis), recurrence (i.e., reappearance of the tumor after treatment in cancer patients), death from any cause, etc. In other words, it represents the survival duration during the observation period when patients do not experience these predefined "events".

SECONDARY OUTCOMES:
2 - year Overall Survival (OS) rate | 2 years
  2 - year Overall Survival (OS) rate: It refers to the proportion of patients who have not died from any cause within the two - year time frame starting from the enrollment. In various cancer clinical trials, regardless of whether the patient's death is caused by cancer itself or other comorbidities (such as infections, failure of other organs, etc.), the time from enrollment to death is defined as OS.
2 - year Distant Metastasis - Free Survival (DMFS) rate | 2 years
  2 - year Distant Metastasis - Free Survival (DMFS) rate: It refers to the proportion of patients whose disease has not developed distant metastasis within the two - year time frame starting from the enrollment. For example, in a clinical study of colorectal cancer, the focus is on the probability of patients surviving without distant organ metastases such as those in the liver and lungs.
2 - year Local Region Recurrence - Free Survival (LRRFS) rate | 2 years
  2 - year Local Region Recurrence - Free Survival (LRRFS) rate: It refers to the proportion of patients who experience no recurrence in the primary tumor site and its surrounding local regions within the two - year time frame starting from enrollment. For instance, in head and neck tumors, the survival probability of patients without tumor recurrence in the primary tumor site of the head and neck, adjacent lymph nodes, and other local regions after treatment represents LRRFS.
Overall Response Rate (ORR) | 2 years
  Overall Response Rate (ORR): Refers to the proportion of patients whose tumor volume reduction meets predetermined criteria and is maintained for a minimum duration. It typically includes cases of complete response (CR, defined as disappearance of all target lesions) and partial response (PR, defined as a ≥30% reduction in the sum of the longest diameters of target lesions), in accordance with RECIST V1.1 criteria.
Duration of Response (DoR) | 2 years
  Duration of Response (DoR): Defined as the time from achieving an objective response (including complete response and partial response) to disease progression or recurrence. For example, in lung cancer targeted therapy, once a patient's tumor shrinkage meets the criteria for partial response following treatment, DoR is the period spanning from this time point until the tumor re-grows or new lesions appear (i.e., disease progression occurs).
Safety(treatment-related toxicity and adverse reactions) | 2 years
  Adverse events (treatment toxicity) will be evaluated using NCI-CTCAE version 5.0. Assessments occur at baseline, during treatment, and through final follow-up to monitor safety profiles.
Patients' Quality of Life | 2 years
  Based on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire ( EORTC QLQ-H&N35) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zeng, Study Chair — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China